CLINICAL TRIAL: NCT00230802
Title: Thyroid Hormone Dose Adjustments During Pregnancy in Women With Primary Hypothyroidism.
Brief Title: Thyroid Hormone Dose Adjustment in Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Erik K. Alexander, Associate Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DK44128 (completed)
Record Dates: First submitted 2005-09-29; First posted 2005-10-03 (Estimated); Results first posted 2016-12-23 (Estimated); Last update posted 2016-12-23 (Estimated); Status verified 2016-10

CONDITIONS: Pregnancy; Hypothyroidism
Keywords: pregnancy; hypothyroidism; levothyroxine
MeSH Terms: conditions — Hypothyroidism | interventions — Thyroxine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 tablet increase (Active Comparator): Patients will increase their current levothyroxine dose by 2 extra tablets per week (~29% increase)
  Interventions: Drug: Anticipatory dose increase of levothyroxine; Drug: levothyroxine
- 3 tablet increase (Active Comparator): Patients will increase their levothyroxine dosage by 3 extra tablets per week (~43%).
  Interventions: Drug: Anticipatory dose increase of levothyroxine; Drug: levothyroxine

INTERVENTIONS:
Drug: Anticipatory dose increase of levothyroxine — as it is know that levothyroxine requirement increases in pregnancy, both study arms will increase levothyroxine dose, though by different amounts.
  Other Names: Levoxyl,; Synthroid,; Unithroid
Drug: levothyroxine — patients will increase levothyroxine dosage by 2 extra tablets of their current dose per week
  Other Names: levoxyl,; synthroid; unithroid
  Arms: 2 tablet increase
Drug: levothyroxine — patients will increase levothyroxine by 3 extra tablets of their current dose per week.
  Other Names: Levoxyl,; Synthroid,; Unithroid
  Arms: 3 tablet increase

SUMMARY:
Our aim is to compare the safety and efficacy of 2 different empiric levothyroxine dose adjustment recommendations to be made at the first confirmation of pregnancy in women with a history of hypothyroidism. Subjects will be women with a prior diagnosis of hypothyroidism who are taking thyroid hormone replacement and who are less than 8 weeks pregnant. Upon confirmation of pregnancy, subjects will be randomized to increase their weekly thyroid hormone dose by either 2 or 3 tablets (28 or 42%). Thyroid function will be evaluated every two weeks in the first 20 weeks and then again at week 30 and post-partum. Primary endpoints will be the proportion of women in each group who remain euthyroid throughout the first trimester and throughout pregnancy.

DETAILED DESCRIPTION:
Our aim is to compare the safety and efficacy of 2 different empiric levothyroxine dose adjustment recommendations to be made at the first confirmation of pregnancy in women with a history of hypothyroidism. Subjects will be women with a prior diagnosis of hypothyroidism who are taking thyroid hormone replacement and who are less than 8 weeks pregnant. Upon confirmation of pregnancy, subjects will be randomized to increase their weekly thyroid hormone dose by either 2 or 3 tablets (28 or 42%). Thyroid function will be evaluated every two weeks in the first 20 weeks and then again at week 30 and post-partum. Primary endpoints will be the proportion of women in each group who remain euthyroid throughout the first trimester and throughout pregnancy

ELIGIBILITY:
Inclusion Criteria:

* women with a prior diagnosis of hypothyroidism, currently receiving levothyroxine therapy
* less than 8 weeks pregnant

Exclusion Criteria:

* cardiac disease, renal failure
* not euthyroid biochemically within 6 months pre-pregnancy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2005-07; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erik Alexander, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Yassa L, Marqusee E, Fawcett R, Alexander EK. Thyroid hormone early adjustment in pregnancy (the THERAPY) trial. J Clin Endocrinol Metab. 2010 Jul;95(7):3234-41. doi: 10.1210/jc.2010-0013. Epub 2010 May 12. PMID 20463094

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 2 Tablet Increase | 3 Tablet Increase
Started | 25 | 23
Completed | 25 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2 Tablet Increase | 3 Tablet Increase | Total
Number analyzed (Participants) | 25 | 23 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 23 | 48
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29 (3) | 28 (5) | 29 (5)
Gender [Count of Participants; unit: Participants]
  Female | 25 | 23 | 48
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 23 | 48

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients in Each Treatment Arm Euthyroid Through Gestation
Description: The proportion of patients in each treatment arm euthyroid through gestation
Time Frame: 9 months
Population: proportion of patients in each treatment arm euthyroid through gestation
Measure: Number; unit: participants
Arm/Group | 2 Tablet Increase | 3 Tablet Increase
Number analyzed (Participants) | 25 | 23
participants | 24 | 21

2. Secondary Outcome: the Participants in Each Arm Who Required Levothyroxine Dose Adjustments (Either Increased or Decreased) Occurred to Maintain a Euthyroid State
Time Frame: 9 months
Measure: Number; unit: participants
Arm/Group | 2 Tablet Increase | 3 Tablet Increase
Number analyzed (Participants) | 25 | 23
participants | 10 | 16

3. Secondary Outcome: Proportion of Subjects With Abnormal Thyroid Stimulating Hormone Values When Following an Every 4 Week Monitoring Schedule During Pregnancy.
Time Frame: 9 months
Measure: Number; unit: participants
Arm/Group | 2 Tablet Increase | 3 Tablet Increase
Number analyzed (Participants) | 25 | 23
participants | 25 | 23

ADVERSE EVENTS:
Arm/Group | 2 Tablet Increase | 3 Tablet Increase
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/23
Other Adverse Events (participants affected / at risk) | 0/25 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No